CLINICAL TRIAL: NCT02855502
Title: Investigation of the Effect of Systemic Steroids on Treatment and Prevention of Recurrent Tracheal Stenosis in Postoperative Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Research Institute of Tuberculosis and Lung Disease, Iran (Other Government)
Responsible Party: Principal Investigator, Shadi Baniasadi, Associate Proffesor, National Research Institute of Tuberculosis and Lung Disease, Iran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: F93162
Record Dates: First submitted 2016-04-17; First posted 2016-08-04 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Tracheal Stenosis
MeSH Terms: conditions — Tracheal Stenosis | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisolone (Active Comparator): dose: 15 mg per day(divided 5 mg TDS) dosage form: tablet duration administration: 30 days
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): placebo given to patient: 3 tablet (divided TDS) dosage form: tablet duration administration: 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone
  Arms: Prednisolone
Drug: Placebo
  Arms: Placebo

SUMMARY:
tracheal stenosis is the result of abnormal wound-healing processes leading to hypertrophic scar formation and obstruction of the airway lumen by excess granulation tissue. This process is progressive so treatment and prevention is essential. Resection-anastomosis of the trachea is becoming the standard of care in many centers and gives the most consistent results in both adult and pediatric patients. But recurrence stenosis, re-granulation and re-inflammation are probable. This study aimed to assess the efficacy of systemic prednisolone on prevention of recurrent tracheal stenosis after surgery.

DETAILED DESCRIPTION:
Tracheal stenosis affects 4-13% of adults and occurs in 1-8% of neonates after prolonged intubation in United States. The causes of adults' tracheal stenosis include trauma, chronic inflammatory diseases, benign neoplasm, malignant neoplasm and collagen vascular diseases. The most common cause of tracheal stenosis continues to be trauma, which can be internal (prolonged endotracheal intubation, tracheostomy, flame, burn injury) or external (neck trauma). Approximately 90% of chronic subglottic stenosis in children and adults results from endotracheal intubation or tracheostomy and about 10% results from other causes.

The resection anastomosis is the most effective treatment to cure this condition. The other treatments are mechanical dilation (dilators, rigid bronchoscopes), stents, laser co2, diode, and cold knife. But they are not as effective as resection anastomosis. Rigid bronchoscopes or dilators may shear the mucosa leading to further damage. Resection of all damaged segments of the airway, approximation and anastomosis of the two intact ends by means of fine synthetic absorbable sutures with minimum tension. Steroids with anti-inflammatory effect widely use as first line therapy for this condition.

Patients who underwent resection anastomosis during 2014-2016 for treatment of post-intubation tracheal stenosis will be included in this study. Systemic prednisolone will be used for treatment and prevention of recurrent tracheal stenosis in post-operative patients. Post-operative patients will divide in two groups, one of them will receive prednisolone and the other will receive placebo for 30 days. The results will be compared by bronchoscopy (FOB or rigid) after 30 days.

ELIGIBILITY:
Inclusion criteria:

1. Post-operative resection anastomosis patients.
2. Age more than 10 years old.
3. no severe tension in surgery by the opinion of surgeon.

Exclusion Criteria:

1. Pregnancy
2. History of significant medical condition not controlled by medicines. Ex: cardiovascular diseases, endocrine impairments and etc.
3. Weight is ≥200% ideal body weight
4. Severe chronic liver disease
5. immunosuppression including HIV+ status, history of bone marrow or solid organ transplantation, current malignancy, neutropenia
6. Fungal systemic infection

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Completely wound healing. | 30 days
  achieved by fiber optic bronchoscopy (FOB) and a surgeon judged that the patients were with out any sign of clinical symptoms of upper respiratory tract stenosis postoperatively and anastomosis site was with out any presence of stenosis (fibrous tissue), granulation tissue formation and inflamed mucosa.

SECONDARY OUTCOMES:
Granulation tissue formation without visible dehiscence | 30 days
  achieved by fiber optic bronchoscopy (FOB) and a surgeon judged about production of fibrotic and excess granulation tissue at the site of anastomosis during FOB.

OTHER OUTCOMES:
inflammation | 30 days
  achieved by fiber optic bronchoscopy (FOB) and surgeon judged the principal etiology of recurrence of an inflammatory process in the anastomosis site which results in development of fibrotic tissue.
Partial and complete dehiscence with or without infection | 30 days
  patients referent hospital emergency, cause of breathing problems and re intubation must needed.

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes